CLINICAL TRIAL: NCT00119106
Title: Study of the Safety and Efficacy of Daily Tenofovir to Prevent HIV Infection Among Injection Drug Users in Bangkok, Thailand
Brief Title: Bangkok Tenofovir Study, an HIV Pre-exposure Prophylaxis Trial, Bangkok, Thailand
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Thailand (Other Government); Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4370
Record Dates: First submitted 2005-07-08; First posted 2005-07-13 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2015-02

CONDITIONS: HIV Infections
Keywords: HIV; Prevention; Tenofovir; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tenofovir disoproxil fumarate (Experimental): Participants in the Tenofovir arm will receive daily oral tenofovir
  Interventions: Drug: Tenofovir disoproxil
- Placebo (Placebo Comparator): Participants in the Placebo are will receive daily oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenofovir disoproxil — Antiretroviral
  Other Names: Tenofovir
  Arms: tenofovir disoproxil fumarate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary goals of this study are to assess the safety and efficacy of daily tenofovir to prevent parenteral HIV infection among injection drug users (IDUs). Assessment of changes in HIV associated risk behaviors, adherence to study drug, and, among IDU who become HIV-infected during the trial, evaluation of HIV viral load set point, CD4 counts, genetic characterization of infecting HIV viruses, and antiretroviral resistance will also be done.

DETAILED DESCRIPTION:
This is a phase II/III, randomized, double-blind, placebo-controlled study of the safety and efficacy of chemoprophylactic tenofovir, administered orally once daily to IDUs. The study will be conducted in Bangkok at 17 BMA Drug Treatment Clinics. Study participants will be randomized (1:1) to receive tenofovir 300 mg or placebo. Participants will be evaluated for adverse events and HIV seroconversion.

Primary endpoints: The primary efficacy endpoint will be measured by rates of HIV seroconversion measured at monthly intervals. The primary safety endpoints will be measured by the frequency of Grade 3 or 4 renal or hepatic function laboratory toxicities or clinical toxicities in blinded tenofovir and placebo arms, as defined by the Gilead-modified NIAID Adult Common Toxicity Tables, and which cannot be directly attributed to a cause other than study medications; and the frequency of adverse clinical events in tenofovir and placebo arms.

Secondary endpoints: Changes in HIV associated risk behaviors will be measured by rates of reported injection drug use and injection drug use frequency during the trial; rates of reported needle sharing; the number of unprotected sexual acts over the course of the trial; number of reported sexual partners over the course of the trial; and proportional use of condoms during sexual intercourse.

Medication adherence will be measured as: rates, by interview and documentation on tenofovir adherence card, of participants taking at least six (86%) of seven daily doses of study drug each of the four weeks preceding the monthly study visit. Differences in virologic and immunologic responses to HIV infection among tenofovir and placebo recipients will be measured by: plasma viral load, measured by quantitative RNA PCR, a predictor of clinical progression of HIV disease; 14 CD4 cell counts will be measured by flow cytometry. Rates and nature of HIV antiretroviral genotypic and phenotypic resistance will be measured. Genetic characteristics of infecting HIV viruses including DNA sequence analysis and antibody binding studies will be conducted.

In phase II, participants will be followed months 0, 1, 2, 3, then 3 monthly with hematology and chemistry tests and laboratory evaluations of renal and hepatic function until 200 person-years of observation are accrued. At that point, a DSMB safety assessment will be conducted. Follow-up of enrolled participants will continue during the DSMB safety assessment. If safety is confirmed, all phase II participants will continue, and additional participants will be enrolled into the phase III portion of the trial. Accrual of the target enrollment of 2,400 IDUs is anticipated to take 48 months.

Participants will choose between two follow-up schedules: monthly (every 4 weeks) or monthly plus daily with directly observed therapy (DOT). During DOT visits clinic staff will witness the participant swallow his/her study medication and clinic staff will initial the participant's tenofovir adherence card. Monthly visits will be the same for both groups and will include an assessment of tenofovir adherence and adverse events, a pill count and collection of unused pills, provision of a new 1 month supply of study medication, pre- and post-test HIV counseling, rapid oral HIV testing, urine pregnancy test (for female participants), HIV risk reduction counseling, and medication adherence counseling. At 3, 6, and every 3 months thereafter monthly procedures will be supplemented with a risk behavior questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Report injection drug use in the 6 months before screening
* Possess a Thai National Identification Card
* Laboratory values as follows within 2 weeks before enrollment:
* HIV oral fluid test non-reactive at screening and pre-enrollment visits
* Hemoglobin 9 gm/dL
* ALT and AST 2.5 x upper limit of normal (ULN)
* Total bilirubin 1.5 mg/dL
* Serum amylase 1.5 x ULN
* Serum phosphorus 2.2 mg/dL
* No evidence of current or chronic Hepatitis B infection by serology
* Calculated creatinine clearance 60 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min = Male: (140 - age in years) x (wt in kg)/72 x (serum creatinine in mg/dL) Female:(140 - age in years) x (wt in kg) x 0.85/72 x (serum creatinine in mg/dL)
* Willing to abstain from sexual intercourse or use effective contraception during the trial (oral, injection, or barrier), for women
* Willing and able to provide informed consent for study participation
* Available and committed to DOT or monthly follow-up for at least 12 months

Exclusion Criteria:

* Clinic physicians will determine if a subject with chronic illness requiring prescription medication can not enroll (medication used for drug treatment is allowed)
* Positive urine pregnancy test
* Breastfeeding
* History of significant renal, liver, or bone disease
* Any other clinical condition or prior therapy that, in the opinion of the clinic physician, would make the subject unsuitable for the study or unable to comply with the dosing requirements
* Concurrent participation in any other HIV prevention trial or drug/vaccine safety trial. AIDSVAX B/E HIV vaccine trial (CDC protocol #2076) participants and Extension Study (CDC protocol #3750) participants may be screened for enrollment in the Bangkok Tenofovir Study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2413 (Actual)
Dates: Start 2005-06; Primary Completion 2013-07 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kachit Choopanya, MD, Principal Investigator — Bangkok Tenofovir Study Group; Michael T Martin, MD, MPH, Study Director — Centers for Disease Control and Prevention; Lynn Paxton, MD, Study Director — Centers for Disease Control and Prevention
Locations (1):
- Thailand Ministry of Public Health - U.S. CDC Collaboration, Nonthaburi, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Concept sheets are reviewed and approved, modified, or declined by research team.
Supporting Information: Study Protocol, ICF
Time Frame: Data available after 2014
Access Criteria: Concept sheets are reviewed and approved, modified, or declined by research team.

REFERENCES:
- [Background] Choopanya K, Martin M, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Kitisin P, Natrujirote P, Kittimunkong S, Chuachoowong R, Gvetadze RJ, McNicholl JM, Paxton LA, Curlin ME, Hendrix CW, Vanichseni S; Bangkok Tenofovir Study Group. Antiretroviral prophylaxis for HIV infection in injecting drug users in Bangkok, Thailand (the Bangkok Tenofovir Study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2013 Jun 15;381(9883):2083-90. doi: 10.1016/S0140-6736(13)61127-7. Epub 2013 Jun 13. PMID 23769234
- [Background] Martin M, Vanichseni S, Suntharasamai P, Sangkum U, Mock PA, Chaipung B, Worrajittanon D, Leethochawalit M, Chiamwongpaet S, Kittimunkong S, Gvetadze RJ, McNicholl JM, Paxton LA, Curlin ME, Holtz TH, Samandari T, Choopanya K; Bangkok Tenofovir Study Group. Factors associated with the uptake of and adherence to HIV pre-exposure prophylaxis in people who have injected drugs: an observational, open-label extension of the Bangkok Tenofovir Study. Lancet HIV. 2017 Feb;4(2):e59-e66. doi: 10.1016/S2352-3018(16)30207-7. Epub 2016 Nov 18. PMID 27866873
- [Background] Martin M, Vanichseni S, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Curlin ME, Na-Pompet S, Warapronmongkholkul A, Kittimunkong S, Gvetadze RJ, McNicholl JM, Paxton LA, Choopanya K; Bangkok Tenofovir Study Group. The impact of adherence to preexposure prophylaxis on the risk of HIV infection among people who inject drugs. AIDS. 2015 Apr 24;29(7):819-24. doi: 10.1097/QAD.0000000000000613. PMID 25985403
- [Background] Martin M, Vanichseni S, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Gvetadze RJ, Kittimunkong S, Curlin ME, Worrajittanon D, McNicholl JM, Paxton LA, Choopanya K; Bangkok Tenofovir Study Group. Risk behaviors and risk factors for HIV infection among participants in the Bangkok tenofovir study, an HIV pre-exposure prophylaxis trial among people who inject drugs. PLoS One. 2014 Mar 25;9(3):e92809. doi: 10.1371/journal.pone.0092809. eCollection 2014. PMID 24667938
- [Background] Vanichseni S, Martin M, Suntharasamai P, Sangkum U, Mock PA, Gvetadze RJ, Curlin ME, Leethochawalit M, Chiamwongpaet S, Chaipung B, McNicholl JM, Paxton LA, Kittimunkong S, Choopanya K. High Mortality Among Non-HIV-Infected People Who Inject Drugs in Bangkok, Thailand, 2005-2012. Am J Public Health. 2015 Jun;105(6):1136-41. doi: 10.2105/AJPH.2014.302473. Epub 2015 Apr 16. PMID 25880964
- [Derived] Parker I, Khalil G, Martin A, Martin M, Vanichseni S, Leelawiwat W, McNicholl J, Hickey A, Garcia-Lerma JG, Choopanya K, Curtis KA. Altered Antibody Responses in Persons Infected with HIV-1 While Using Preexposure Prophylaxis. AIDS Res Hum Retroviruses. 2021 Mar;37(3):189-195. doi: 10.1089/AID.2020.0137. Epub 2020 Dec 9. PMID 33126825
- [Derived] Suntharasamai P, Martin M, Choopanya K, Vanichseni S, Sangkum U, Tararut P, Leelawiwat W, Anekvorapong R, Mock PA, Cherdtrakulkiat T, Leethochawalit M, Chiamwongpaet S, Gvetadze RJ, McNicholl JM, Paxton LA, Kittimunkong S, Curlin ME. Assessment of Oral Fluid HIV Test Performance in an HIV Pre-Exposure Prophylaxis Trial in Bangkok, Thailand. PLoS One. 2015 Dec 30;10(12):e0145859. doi: 10.1371/journal.pone.0145859. eCollection 2015. PMID 26717405
- [Derived] Martin M, Vanichseni S, Suntharasamai P, Sangkum U, Mock PA, Gvetadze RJ, Curlin ME, Leethochawalit M, Chiamwongpaet S, Cherdtrakulkiat T, Anekvorapong R, Leelawiwat W, Chantharojwong N, McNicholl JM, Paxton LA, Kittimunkong S, Choopanya K; Bangkok Tenofovir Study Group. Renal function of participants in the Bangkok tenofovir study--Thailand, 2005-2012. Clin Infect Dis. 2014 Sep 1;59(5):716-24. doi: 10.1093/cid/ciu355. Epub 2014 May 14. PMID 24829212
- [Derived] Martin M, Vanichseni S, Suntharasamai P, Sangkum U, Chuachoowong R, Mock PA, Leethochawalit M, Chiamwongpaet S, Kittimunkong S, van Griensven F, McNicholl JM, Paxton L, Choopanya K; Bangkok Tenofovir Study Group. Enrollment characteristics and risk behaviors of injection drug users participating in the Bangkok Tenofovir Study, Thailand. PLoS One. 2011;6(9):e25127. doi: 10.1371/journal.pone.0025127. Epub 2011 Sep 28. PMID 21969870

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenofovir: Tenofovir
  Tenofovir
- Placebo: Placebo
  Tenofovir
Period: Overall Study
Arm/Group | Tenofovir | Placebo
Started | 1204 | 1209 (2 participants later found to be HIV infected at baseline. Therefore 1207 in mITT analysis)
Completed | 1025 | 1031
Not Completed | 179 | 178
Not completed — HIV infected at baseline | 179 | 178

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir | Placebo | Total
Number analyzed (Participants) | 1204 | 1207 | 2411
Age, Continuous [Median (Standard Deviation); unit: years] | 31 (8) | 31 (8) | 31 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 241 | 487
  Male | 958 | 966 | 1924
Region of Enrollment [Number; unit: participants]
  Thailand | 1204 | 1207 | 2411

OUTCOME MEASURES:

1. Primary Outcome: Rates of HIV Seroconversion
Description: Kaplan Meier survival curve.
Time Frame: From date of randomization until the date of first documented seroconversion or date of death from any cause, whichever came first, assessed for an average of 4.0 years, with a maximum duration of 6.9 years
Measure: Number; unit: Infections/ 100 person-years
Arm/Group | Tenofovir | Placebo
Number analyzed (Participants) | 1204 | 1209
Infections/ 100 person-years | 17 | 33

2. Primary Outcome: Renal Toxicity
Description: Number of Participants with Grade 3 or 4 Renal Laboratory Toxicities
Time Frame: Blood tested for creatinine level at enrollment and every 3 months, up to 6.9 years
Population: creatinine clearance measured in all participants every 3 months
Measure: Number; unit: participants
Arm/Group | Tenofovir | Placebo
Number analyzed (Participants) | 1204 | 1209
participants | 3 | 3

3. Primary Outcome: Adverse Events
Description: Number of Participants with adverse clinical events in tenofovir and placebo arms
Time Frame: Up to 6.9 years
Measure: Number; unit: participants
Arm/Group | Tenofovir | Placebo
Number analyzed (Participants) | 1204 | 1209
participants | 1098 | 1083

4. Secondary Outcome: Number of Participants Reporting Injecting and Sharing Needles
Description: Number of Participants reporting injecting and sharing needles:
  Assessed injecting and sharing at baseline and every 3 months during follow-up. We used GEE to determine if there was a significant decline in injecting and sharing.
Time Frame: Participants were asked about injecting and needle sharing behaviors at enrollment and every 3 month visit, up to 6.9 years
Measure: Number; unit: participants
Arm/Group | Tenofovir | Placebo
Number analyzed (Participants) | 1204 | 1207
participants | 58 | 59

5. Secondary Outcome: Adherence to Study Drug/Placebo
Description: Mean number of days that participants took study drug based on study drug diaries by study group.
Time Frame: Participants were asked about adherence at 3 month visits, up to 6.9 years.
Population: All participants
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tenofovir | Placebo
Number analyzed (Participants) | 1204 | 1207
days | 84 (23) | 84 (23)

6. Secondary Outcome: HIV Viral Load Copies/mL Measured at First Positive HIV Test Result by Group
Description: Plasma HIV RNA concentrations.
Time Frame: Among people who seroconverted, viral load was measured at month 1, 2, and every 4 months after HIV seroconversion
Population: Participants who seroconverted during follow-up.
Measure: Mean (Standard Deviation); unit: Copies/mL
Groups:
- Tenofovir: Received tenofovir
- Placebo: Received placebo
Arm/Group | Tenofovir | Placebo
Number analyzed (Participants) | 33 | 17
Copies/mL | 929829 (2272690) | 120061 (222612)

7. Secondary Outcome: Number Participants Who Reported More Than One Sexual Partner at Baseline
Description: Number of participants
Time Frame: At enrolment
Measure: Count of Participants; unit: Participants
Groups:
- Tenofovir Group: Tenofovir participants
- Placebo Group: Placebo recipients
Arm/Group | Tenofovir Group | Placebo Group
Number analyzed (Participants) | 1204 | 1209
Participants | 251 | 271

8. Secondary Outcome: Number of Participants With Tenofovir-associated Resistance Mutations.
Description: Measure tenofovir associated resistance mutations (ie, K65R and K70E) in amplified viral RNA specimens from HIV-positive participants in the placebo and tenofovir groups.
Time Frame: Specimens collected at the time of HIV seroconversion
Measure: Count of Participants; unit: Participants
Groups:
- Tenofovir; Placebo: Participants
Arm/Group | Tenofovir | Placebo
Number analyzed (Participants) | 14 | 29
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events from the date the participant enrolled and started study drug until the participant completed follow-up, a maximum of 6.9 years.
Arm/Group | Tenofovir | Placebo
All-Cause Mortality (participants affected / at risk) | 49/1204 | 58/1209
Serious Adverse Events (participants affected / at risk) | 227/1204 | 246/1209
Other Adverse Events (participants affected / at risk) | 1098/1204 | 1083/1209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir (N=1204) | Placebo (N=1209)
Any serious adverse event (Investigations) | 227 (340) | 246 (375)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir (N=1204) | Placebo (N=1209)
AE (Investigations) | 1098 (10965) | 1083 (11550) — Other adverse events
Renal toxicity (Renal and urinary disorders) | 3 (4) | 3 (3) — NIH Grade 3 or 4

LIMITATIONS AND CAVEATS:
Participants could have under-reported stigmatised behaviours such as injecting drugs.30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No